CLINICAL TRIAL: NCT05369416
Title: Renal Metabolism in Salt-sensitive Human Blood Pressure
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Srividya Kidambi, MD, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PRO00037003
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Hypertension
Keywords: hypertension; high blood pressure; salt
MeSH Terms: conditions — Hypertension | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Masking Description: We are using a crossover design of low-sodium and high-sodium diets of 2 week duration each.
  Both diets consecutively given to each subject recruited in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low sodium diet (Active Comparator): -Subjects will be randomized to start a low sodium diet (1200 mg/day) for two weeks (this will be followed by a high sodium diet - crossover design)
  Interventions: Other: Low sodium diet
- high sodium diet (Active Comparator): -Subjects will be randomized to start a high sodium diet (4200 mg/day) for two weeks (this will be followed by a low sodium diet - crossover design)
  Interventions: Other: high sodium diet

INTERVENTIONS:
Other: Low sodium diet — Subjects will be started on a low sodium (food will be provided) for two weeks.
  Arms: Low sodium diet
Other: high sodium diet — Subjects will be started on high sodium diet (regular diet supplemented with salt tablets to reach a daily intake of > 4200 mg/Day) for two weeks.
  Arms: high sodium diet

SUMMARY:
Salt sensitive hypertension is a significant health problem worldwide and a primary modifiable risk factor for renal, cardiovascular, and cerebrovascular diseases. Yet, the underlying mechanisms remain poorly understood.

The proposed study determines how renal oxygenation and substrate metabolism differs between individuals with and without salt sensitivity, with the ultimate goal of identifying mechanisms, diagnostic criteria, and treatment strategies for salt sensitive hypertension.

DETAILED DESCRIPTION:
Seventy subjects will be enrolled and randomized to start either a low sodium diet (1200 mg/day) or high sodium diet (>4200 mg/day) for two weeks. After completion of two weeks, subjects will be switched to the 'other' diet for two weeks after a one-week wash-out. During the screening visit, subject's daily sodium intake will be assessed using multiple methods and further dietary information will be collected to prepare customized low sodium meals. During low sodium diet period, subjects will be supplied with food and will be asked to keep food logs. At the end of two-week period, the study activities described below will be carried out including BOLD MRI imaging along with imaging techniques to assess renal oxygenation levels and perfusion. During high sodium diet period, subjects will be either supplemented with sodium chloride tablets or high sodium foods to achieve a daily sodium intake above 4200 mg/day. If subjects already consume over 4200 mg/day of sodium, no changes will be made to their diet and assessment of oxygenation (BOLD MRI) and perfusion will take place after two weeks.

At the end of high sodium diet, 18 subjects will have renal vein sampling performed (this will be equally divided between salt-sensitive and salt-insensitive subjects and per subject preference as all may not want to have renal vein sampling). Subjects will be classified into salt sensitive or insensitive at the end of low sodium diet period based on BP response for further data analyses.

ELIGIBILITY:
Inclusion Criteria:

* English speaking subjects
* With a spectrum of BPs, ranging from those with Elevated BP through Stage 1 HTN, as defined by the 2017 ACC/AHA HTN guidelines

Exclusion Criteria:

* Non-English speakers
* BP ≤120/80 & ≥ 140/90 mmHg
* H/o diabetes, congestive heart failure, cirrhosis of the liver, hypokalemia & other
* electrolyte disturbances
* H/o kidney disease
* Use of glucocorticoids
* Pregnant or nursing mothers
* Presence of bleeding disorders
* Use of anti-platelet and anticoagulant agents such as clopidogrel, aspirin, dabigatran, rivaroxaban etc
* Daily sodium intake ≥ 6000 mg/day
* Presence of pacemaker or other metallic implants
* Allergy to iodinated contrast
* Allergy to shellfish
* Claustrophobia

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2030-01-30 (Estimated); Study Completion 2030-01-30 (Estimated)

PRIMARY OUTCOMES:
Changes in renal regional tissue oxygenation in response to salt intake and salt sensitivity | 6 weeks
  70 subjects (~50% women, ~50% AA) will be recruited and salt sensitivity will be determined (defined as ≥8 mmHg decrease in systolic BP on a low Na+ diet). BOLD-MRI and MRI with arterial spin labeling (MRI-ASL) will be performed to assess renal regional tissue oxygenation and perfusion at baseline and after high and low Na+ diets.

SECONDARY OUTCOMES:
Changes in renal metabolites in response to a high sodium diet among individuals who are salt-sensitive versus insensitive | 6 weeks
  In a sub-sample (n=18), metabolomic analysis on peripheral blood and urine samples at baseline and at the end of both diet periods will be performed. These measures will include circulating and urine levels of ketones, acetate and lactate. In addition, peripheral arterial and renal vein samples will be obtained after high Na+ diet period for metabolomic analysis. The concurrent sampling of urine, arterial, and renal venous blood and metabolomics analyses will allow us to comprehensively assess renal uptake and release of metabolites in humans for the first time.

CONTACTS AND LOCATIONS:
Overall Officials: Srividya Kidambi, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin /Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No